CLINICAL TRIAL: NCT04310020
Title: A Pilot Study of Hypofractionated Radiotherapy Followed by Atezolizumab Consolidation in Stage II or III NSCLC Patients With Borderline Performance Status
Brief Title: Study of Radiation Therapy Followed by Atezolizumab in Stage II or III Non-small Cell Lung Cancer Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-01543; NCI-2020-01543 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1933 (Other: SWOG); S1933 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2020-03-16; First posted 2020-03-17 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-10

CONDITIONS: Lung Non-Small Cell Carcinoma; Stage II Lung Cancer AJCC v8; Stage III Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — atezolizumab; Specimen Handling; Radiation Dose Hypofractionation; Radiation; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (hypofractionated radiation therapy, atezolizumab) (Experimental): RADIATION THERAPY: Patients undergo hypofractionated radiation therapy 5 days per week over 3 weeks for 15 fractions in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients receive atezolizumab IV over 30-60 minutes on day 1 of each cycle. Cycles repeat every 21 days for up to 12 months (maximum of 17 cycles) in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan and may undergo MRI throughout the study, as well as blood sample collection on study.
  Interventions: Drug: Atezolizumab; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Radiation: Hypofractionated Radiation Therapy; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG 7446; RG-7446; RG7446; RO 5541267; RO-5541267; RO5541267; Tecentriq
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Radiation: Hypofractionated Radiation Therapy — Undergo hypofractionated radiation therapy
  Other Names: Hypofractionated; Hypofractionated Radiotherapy; hypofractionation; Radiation, Hypofractionated
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI

SUMMARY:
This phase II trial studies the side effects of radiation therapy followed by atezolizumab in treating patients with stage II or III non-small cell lung cancer. Hypofractionated radiation therapy delivers higher doses of radiation therapy over a shorter period of time and may kill more cancer cells and have fewer side effects. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. The purpose of this study is to test the safety and effectiveness of radiation therapy followed by atezolizumab and find out what side effects, if any, it has on patient's non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the rate of grade 3-5 treatment-related adverse events (TRAEs) in patients who are not candidates for surgery or concurrent chemoradiation and who have either performance status 0-2 and stage II or performance status 2 and stage III non-small cell lung cancer (NSCLC), treated with hypofractionated thoracic radiotherapy followed by atezolizumab.

SECONDARY OBJECTIVES:

I. To evaluate response rate (confirmed and unconfirmed, complete and partial by Response Evaluation Criteria in Solid Tumors [RECIST] 1.1) from Registration Step 2 in the subset of patients with measurable disease.

II. To evaluate response rate (confirmed and unconfirmed, complete and partial by RECIST 1.1) during radiation therapy in the subset of patients with measurable disease.

III. To evaluate progression free survival (PFS) from Registration Step 2 by RECIST 1.1.

IV. To evaluate overall survival (OS) from Registration Step 2. V. To evaluate the frequency and severity of toxicities.

ADDITIONAL OBJECTIVE:

I. To bank blood and archival tissue for future research.

OUTLINE:

RADIATION THERAPY: Patients undergo hypofractionated radiation therapy 5 days per week over 3 weeks for 15 fractions in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION: Patients receive atezolizumab intravenously (IV) over 30-60 minutes on day 1 of each cycle. Cycles repeat every 21 days for up to 12 months (maximum of 17 cycles) in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) scan and may undergo magnetic resonance imaging (MRI) throughout the study, as well as blood sample collection on study.

After completion of study treatment, patients are followed up at 6 weeks, every 12 months for the 1 year, then every 6 months until 3 years after study start.

ELIGIBILITY:
Inclusion Criteria:

* REGISTRATION STEP 1: Participants must have pathologic (cytological or histological) proof of non-small cell lung cancer (NSCLC)
* REGISTRATION STEP 1: Participants must have stage III NSCLC with Zubrod performance status of 2 or stage II NSCLC with Zubrod performance status of 0-2
* REGISTRATION STEP 1: Participants must not be candidates for surgical resection in the opinion of the treating investigator. Participants whose disease was previously resected must have experienced local or regional recurrence at least 12 months after resection
* REGISTRATION STEP 1: Participants must not be candidates for concurrent chemoradiation in the opinion of the treating investigator
* REGISTRATION STEP 1: Participants must have measurable or non-measurable disease documented by CT or MRI. Measurable disease must be assessed within 28 days prior to Registration Step 1. Non-measurable disease must be assessed within 42 days prior to Step 1 registration. The CT from a combined positron emission tomography (PET)/CT may be used only if it is of diagnostic quality. All known sites of disease must be assessed and documented on the Baseline Tumor Assessment Form (RECIST 1.1)
* REGISTRATION STEP 1: Participants must have an MRI or CT scan of the brain with contrast within 28 days prior to Registration Step 1
* REGISTRATION STEP 1: Participants' disease must fit within the radiation constraints in the opinion of a local radiation oncologist
* REGISTRATION STEP 1: Participants may have received prior treatment for their lung cancer, including surgery, chemotherapy, targeted agents, and/or radiation treatment. At least 12 months must have elapsed since last treatment
* REGISTRATION STEP 1: Participants may have had prior radiation therapy as long as the irradiated area does not overlap with the radiation field targeted for this study
* REGISTRATION STEP 1: Participants must have recovered from any adverse effects of prior major surgery to the satisfaction of the treating physician. Biopsies and central IV access placement are not considered major surgery
* REGISTRATION STEP 1: Absolute neutrophil count (ANC) >= 1500/mcl (obtained within 28 days prior to Registration Step 1)
* REGISTRATION STEP 1: Platelet count >= 100,000/mcl (obtained within 28 days prior to Registration Step 1)
* REGISTRATION STEP 1: Hemoglobin >= 9 grams/dL (obtained within 28 days prior to Registration Step 1)
* REGISTRATION STEP 1: Total bilirubin =< 1.5 x institutional upper limit of normal (IULN) (obtained within 28 days prior to Registration Step 1)
* REGISTRATION STEP 1: Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x IULN (obtained within 28 days prior to Registration Step 1)
* REGISTRATION STEP 1: Serum creatinine =< 1.5 x IULN OR measured or calculated creatinine clearance >= 40 mL/min (obtained within 28 days prior to Registration Step 1)
* REGISTRATION STEP 1: Participants must have percent predicted diffusing capacity of the lungs for carbon monoxide (DLCO) of at least 40% documented within 90 days prior to Registration Step 1
* REGISTRATION STEP 1: Patient must not have had a prior history of interstitial lung disease or > grade 2 (Common Terminology Criteria for Adverse Events [CTCAE] version 5) pneumonitis
* REGISTRATION STEP 1: Participants must not have active autoimmune disease requiring therapy within the past 6 months
* REGISTRATION STEP 1: Participants must not have an active infection requiring therapy
* REGISTRATION STEP 1: Participants must be ≥ 18 years old
* REGISTRATION STEP 1: Participants must not be pregnant or nursing because atezolizumab has not been studied in pregnant or nursing women and the mechanism of action is expected to cause fetal harm. Women/men of reproductive potential must have agreed to use an effective contraceptive method while on protocol treatment and for five months after last dose of atezolizumab. A woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months. In addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation. However, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures
* REGISTRATION STEP 1: Participants with known human immunodeficiency virus (HIV) infection must be on effective anti-retroviral therapy and must have undetectable viral load at their most recent viral load test and within 6 months prior to Registration Step 1
* REGISTRATION STEP 1: Patient must be tested for hepatitis B within 28 days prior to Registration Step 1. Patient must not have active (chronic or acute) hepatitis B virus (HBV) infection. Patients may have past or resolved HBV infection. Active HBV is defined as having a positive hepatitis B surface antigen (HBsAg) test. Past or resolved HBV is defined as having a negative HBsAG test and a positive total hepatitis B core antibody (HBcAb) test
* REGISTRATION STEP 1: Patients must not have active hepatitis C virus (HCV) infection. Active HCV is defined as having a positive HCV antibody test followed by a positive HCV ribonucleic acid (RNA) test. Patient must have an HCV antibody test within 28 days prior to Registration Step 1. If the HCV antibody test is positive, the patient must also have an HCV quantitative RNA test within 28 days prior to Registration Step 1
* REGISTRATION STEP 1: No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for three years. Participants with localized prostate cancer who are being followed by an active surveillance program are also eligible
* REGISTRATION STEP 1: Participants must be offered optional participation in banking of specimens for future research
* REGISTRATION STEP 1: Participants must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* REGISTRATION STEP 1: As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system
* REGISTRATION STEP 2: Participants must be registered to Step 2 within 42 days after completion of radiation treatment. Participants must have received at least 44 Gy of radiation treatment
* REGISTRATION STEP 2: Participants must have no evidence of progression per RECIST 1.1 on CT scan of the chest, abdomen, and pelvis performed between 2 and 5 weeks after completion of radiation therapy
* REGISTRATION STEP 2: Any toxicities from radiation therapy must have resolved to < grade 2
* REGISTRATION STEP 2: ANC >= 1.5 x 10^3/uL (obtained within 28 days prior to Registration Step 2)
* REGISTRATION STEP 2: Platelet count >= 100 x 10^3/uL (obtained within 28 days prior to Registration Step 2)
* REGISTRATION STEP 2: Hemoglobin >= 9 grams/dL (obtained within 28 days prior to Registration Step 2)
* REGISTRATION STEP 2: Total bilirubin =< 1.5 x institutional upper limit of normal (IULN) (obtained within 28 days prior to Registration Step 2)
* REGISTRATION STEP 2: AST and ALT =< 2.5 x IULN (obtained within 28 days prior to Registration Step 2)
* REGISTRATION STEP 2: Serum creatinine =< 1.5 x IULN OR measured or calculated creatinine clearance >= 40 mL/min (obtained within 28 days prior to Registration Step 2)
* REGISTRATION STEP 2: Participants must not have received steroids in doses of more than prednisone 10 mg daily or equivalent within 14 days prior to Registration Step 2
* REGISTRATION STEP 2: Participants must not have received a live vaccine within 28 days prior to Registration Step 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2021-01-13 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Rate of grade 3-5 adverse events | From baseline, until 180 days from Step 2 registration
  Individual toxicities with possible, probable or likely attribution to treatment along with the overall rate of grade 3, 4 or 5 toxicities attributable to treatment will be summarized.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 3 years
  Individual toxicities with possible, probable or likely attribution to treatment along with the overall rate of grade 3, 4 or 5 toxicities attributable to treatment will be summarized.
Response rate (confirmed and unconfirmed, complete and partial by Response Evaluation Criteria in Solid Tumors [RECIST] 1.1) in the subset of patients with measurable disease (Registration Step 2) | After atezolizumab treatment
  Binary endpoints will be summarized as proportions with 95% Clopper-Pearson confidence intervals.
Response rate (confirmed and unconfirmed, complete and partial by RECIST 1.1) in the subset of patients with measurable disease (Registration Step 1) | During radiation therapy
  Binary endpoints will be summarized as proportions with 95% Clopper-Pearson confidence intervals.
Progression-free survival | From date of Step 2 registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause, assessed up to 3 years
  Estimated using the method of Kaplan-Meier. 95% confidence for the medians will be constructed using the method of Brookmeyer-Crowley.
Overall survival | From date of Step 2 registration to date of death due to any cause, assessed up to 3 years
  Estimated using the method of Kaplan-Meier. 95% confidence for the medians will be constructed using the method of Brookmeyer-Crowley.

CONTACTS AND LOCATIONS:
Overall Officials: Raid Aljumaily, Principal Investigator — SWOG Cancer Research Network
Locations (172):
- United States (172):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - AdventHealth Porter, Denver, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Augusta University Medical Center, Augusta, Georgia
  - CTCA at Southeastern Regional Medical Center, Newnan, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Saint Mary's Hospital, Centralia, Illinois
  - Jesse Brown Veterans Affairs Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Saint Joseph Hospital, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Beverly Hospital, Beverly, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Lahey Medical Center-Peabody, Peabody, Massachusetts
  - Beth Israel Deaconess Medical Center/Winchester Center for Cancer Care, Winchester, Massachusetts
  - Henry Ford Health Providence Novi Hospital, Novi, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Fairview Southdale Hospital, Edina, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Center at UPMC Horizon, Farrell, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Hillman Cancer Center in Greenville/UPMC Horizon, Greenville, Pennsylvania
  - UPMC Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center - New Castle, New Castle, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Cancer Center-Washington, Washington, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern Simmons Cancer Center - RedBird, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Ascension Saint Elizabeth Hospital, Appleton, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Ascension Calumet Hospital, Chilton, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Franklin, Franklin, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Saint Joseph Campus, Milwaukee, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Ascension Saint Francis Hospital, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Ascension Mercy Hospital, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Ascension Medical Group Southeast Wisconsin - Mayfair Road, Wauwatosa, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm